CLINICAL TRIAL: NCT04572308
Title: Cell Therapy for CD7 Positive T-cell Acute Lymphoblastic Leukemia and Lymphoblastic Lymphoma Using CD7-Specific CAR-T Cells
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Hebei Senlang Biotechnology Inc., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CD7 CAR-T for T-ALL/T-LBL
Record Dates: First submitted 2020-09-27; First posted 2020-10-01 (Actual); Last update posted 2021-06-29 (Actual); Status verified 2021-06

CONDITIONS: T-cell Acute Lymphoblastic Leukemia/Lymphoma
Keywords: T-ALL，T-LBL , CD7，CAR-T
MeSH Terms: conditions — Precursor T-Cell Lymphoblastic Leukemia-Lymphoma; Lymphoma

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- CD7 CAR-T (Experimental): Patients will be treated with CD7 CAR-T cells
  Interventions: Biological: CD7 CAR-T

INTERVENTIONS:
Biological: CD7 CAR-T — Patients will be treated with CD7 CAR-T cells
  Biological: CD7 CAR-T; Drug: Cyclophosphamide,Fludarabine; Procedure: Leukapheresis;

SUMMARY:
This is an open, single-arm, clinical study to evaluate efficacy and safety of anti CD7 CAR-T cell in the treatment of relapsed or refractory T-cell acute lymphoblastic leukemia (T-ALL) and lymphoblastic lymphoma (TLBL).

DETAILED DESCRIPTION:
The CARs consist of an anti-CD7 single-chain variable fragment（scFv）, a portion of the human CD137（4-1BB） molecule, and the intracellular component of the human CD3ζ molecule. Prior to CAR-T cell infusion, the patients will be subjected to preconditioning treatment. After CAR-T cell infusion, the patients will be evaluated for adverse reactions and efficacy.

The Main research objectives:

To evaluate the safety and efficacy of CD7 CAR-T cells in patients with relapsed or refractory T-ALL/LBL

The Secondary research objectives:

To investigate the cytokinetic characteristics of CD7 CAR-T cells in patients with relapsed or refractory T-ALL/LBL

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosis of refractory or relapsed T-cell acute lymphoblastic leukemia (T-ALL) or lymphoblastic lymphoma (T-LBL) according to the NCCN 2019.V2 Guideline. Refractory T-ALL is defined as a patient who has failed to achieve complete remission after induction therapy. Relapsed T-ALL is defined as the reappearance of blasts (5%) in either peripheral blood or bone marrow. Patients whose tumor burden >5% blasts, or who have persistent positive minimal residual disease (MRD), or have reappearance of extramedullary lesions are also considered eligible.
2. CD7-positive tumor (≥70% CD7 positive blasts by flow cytometry or immunohistochemistry (tissue) assessed by a CLIA certified Flow Cytometry/Pathology laboratory). tumors burden >5%,or MRD+， or new extramedullary lesions reappeared.
3. Life expectancy greater than 12 weeks
4. KPS or Lansky score≥60
5. HGB≥70g/L
6. oxygen saturation of blood>90%
7. Total bilirubin (TBil)≤3 × upper limit normal, aspartate aminotransferase (AST) and alanine aminotransferase (ALT) ≤ 5×upper limit of normal
8. Informed consent explained to, understood by and signed by patient/guardian.

Exclusion Criteria:

1. Any of the following cardiac criteria: Atrial fibrillation/flutter; Myocardial infarction within the last 12 months; Prolonged QT syndrome or secondary prolonged QT, per investigator discretion. Cardiac echocardiography with LVSF (left ventricular shortening fraction)<30% or LVEF(left ventricular ejection fraction)<50%; or clinically significant pericardial effusion. Cardiac dysfunction NYHA(New York Heart Association) III or IV (Confirmation of absence of these conditions on echocardiogram within 12 months of treatment)
2. Has an active GvHD;
3. Has a history of severe pulmonary function damaging;
4. With other tumors which is/are in advanced malignant and has/have systemic metastasis;
5. Severe or persistent infection that cannot be effectively controlled；
6. Presence of severe autoimmune diseases or immunodeficiency disease;
7. Patients with active hepatitis B or hepatitis C([HBVDNA+]or [HCVRNA+]);
8. Patients with HIV infection or syphilis infection;
9. Has a history of serious allergies to biological products (including antibiotics);
10. Clinically significant viral infection or uncontrolled viral reactivation of EBV(Epstein-Barr virus), CMV(cytomegalovirus), ADV(adenovirus), BK-virus, or HHV(human herpesvirus)-6.
11. Presence of any symtomatic CNS disorder such as an uncontrolled seizure disorder, cerebrovascular ischemia/hemorrhage, dementia, cerebellar disease, or any autoimmune disease with CNS involvement;
12. Received allogeneic hematopoietic stem cell transplantation within 6 months;
13. Being pregnant and lactating or having pregnancy within 12 months;
14. Any situations that the researchers believe will increase the risks for the subject or affect the results of the study.

Ages: 2 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2020-10-01 (Actual); Primary Completion 2021-05-30 (Actual); Study Completion 2021-05-30 (Actual)

PRIMARY OUTCOMES:
Safety: Incidence and severity of adverse events | First 1 month post CAR-T cells infusion
  To evaluate the possible adverse events occurred within the first one month after CD7 CAR-T infusion, including the incidence and severity of symptoms such as cytokine release syndrome and neurotoxicity
Efficacy: Remission Rate | 3 months post CAR-T cells infusion
  Remission Rate including complete remission(CR)、CR with incomplete blood count recovery(CRi)、partial remission(PR), No remission(NR), overall remission (OR)

SECONDARY OUTCOMES:
duration of response (DOR) | 24 months post CAR-T cells infusion
  duration of response (DOR)
Efficacy: progression-free survival (PFS) | 24 months post CAR-T cells infusion
  progression-free survival (PFS) time
CAR-T proliferation | 3 months post CAR-T cells infusion
  the copy number of CD7 CAR- T cells in the genomes of PBMC by qPCR method
CAR-T proliferation | 3 months post CAR-T cells infusion
  percentage of CD7 CAR- T cells measured by flow cytometry method
Cytokine release | First 1 month post CAR-T cells infusion
  Cytokine( IL-6,IL-10,IFN-γ,TNF-α ) concentration (pg/mL) by flow cytometry method
Pharmacokinetics (PK) indicators: | Long time
  the peak concentration of Senl-T7 CAR-T cells amplified in the peripheral blood (Cmax, detected by flow cytometry and qPCR); the time taken to reach the peak concentration (Tmax), and the persistent time of the Senl-T7 CAR-T cells in vivo in patients;
Pharmacodynamic (PD) indicators: | First 1 month post CAR-T cells infusion
  the pharmacodynamic change in the clearance of peripheral blood CD7+ cells and the release of the cytokines at each observation time point

CONTACTS AND LOCATIONS:
Locations (1):
- Hebei yanda Ludaopei Hospital, Yanda, Hebei, China

REFERENCES:
- [Derived] Velasquez MP. Allogeneic CD7-CAR T cells to bridge the gap? Transplant Cell Ther. 2023 Mar;29(3):139-140. doi: 10.1016/j.jtct.2023.02.006. No abstract available. PMID 36858787